CLINICAL TRIAL: NCT05635136
Title: Histopathological Analysis of Renal Biopsies With Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings in Kidney Transplant Recipients
Brief Title: Histopathological Analysis of Renal Biopsies With Dynamic Full-field Optical Coherence Tomography, a Comparison to Conventional Histopathological Findings in Kidney Transplant Recipients (HARBOR)
Acronym: HARBOR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier William Morey - Chalon sur Saône (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Other Study IDs: HARBOR
Record Dates: First submitted 2022-11-14; First posted 2022-12-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Tomography, Optical Coherence; Kidney Transplantation
Keywords: Kidney Transplantation; Kidney Biopsy; Full-field Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The DIVAT cohort: patient > 18 years of age who received renal transplant are registered in the DIVAT cohort (standing for computerized and validated data in transplantation, "Données Informatisées VAlidées Transplantation"). It comprises more than 300 clinical and biological parameters collected at the time of transplant, at 3 months, 6 months and at each anniversary of the transplant. The DIVAT cohort and network is accredited by the CNIL (standing for "Commission Nationale de l'Informatique et des Libertés")
  Interventions: Other: Dynamic full-field optical coherence tomography analysis of kidney transplant biopsy

INTERVENTIONS:
Other: Dynamic full-field optical coherence tomography analysis of kidney transplant biopsy — Dynamic full-field optical coherence tomography analysis of kidney transplant biopsy before conventional histopathological analysis

SUMMARY:
Banff classification stands as gold standard and international consensus for the identification, diagnosis and categorization of renal allograft pathology. In addition to multiple revision dedicated to the clarification and refinement of these diagnostic categories, a special attention is now dedicated to the development of automated protocols serving the use of artificial intelligence in digital pathology. To be integrated in the actual early post-transplant monitoring procedure, such original approach is considered to match various growing expectations of clinicians and pathologists regarding the future of transplant nephropathology : decrease inter-observer variability, reduce human errors and limit time-consuming analysis of kidney biopsy. Among these, an accelerated reading and access to Banff diagnostic criteria could help initiating both appropriate and immediate treatment to improve graft survival in kidney transplant recipients. Yet conventional histopathology still requires the preparation of a paraffin block, sections as well as subsequent colorations that altogether delay the final pathological diagnosis and urge the need for additional diagnostic modalities. Designed to overcome this critical limitation, the HARBOR study intends to test the performance of direct histopathological examination of fresh kidney biopsy with full-field optical coherence tomography for the identification of Banff elemental lesions and diagnostic categories.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years of age who received renal transplant registered in the DIVAT cohort with kidney biopsy between start study date and primary completion date

Exclusion Criteria:

* inability to perform dynamic full-field optical coherence tomography observation at the moment of kidney biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient > 18 years of age who received renal transplant are registered in the DIVAT cohort. It comprises more than 300 clinical and biological parameters collected at the time of transplant, at 3 months, 6 months and at each anniversary of the transplant. The DIVAT cohort and network is accredited by the CNIL (Commission Nationale de l'Informatique et des Libertés)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Banff lesion scores based on dynamic full-field optical coherence tomography measurement | Outcome measure is assessed 15 days following kidney transplant biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify and score the usual Banff lesions comprising interstitial inflammation, tubulitis, intimal arteritis, glomerulitis, peritubular capillaritis, interstitial fibrosis, tubular atrophy, vascular fibrous intimal thickening, glomerular basement membrane double contours, mesangial matrix expansion, arteriolar hyalinosis, hyaline arteriolar thickening, total inflammation and inflammation in the area of both interstitial fibrosis and tubular atrophy.
  Note that the the Banff scoring system has three grades for each lesion : from mild (1) to moderate (2) and severe (3). In each case, the higher the score the worse the outcome, according to the 2018 Reference Guide to the Banff Classification of Renal Allograft Pathology

SECONDARY OUTCOMES:
Banff diagnostic categories based on dynamic full-field optical coherence tomography measurement | Outcome measure is assessed 15 days following kidney transplant biopsy
  Provide a better understanding of the ability of dynamic full-field optical coherence tomography to identify the usual Banff diagnostic categories comprising normal biopsy (or biopsy with nonspecific changes), biopsy with antibody-mediated changes, biopsy considered borderline or suspicious for acute T cell-mediated rejection, biopsy with T cell-mediated rejection, biopsy with both interstitial fibrosis and tubular atrophy, biopsy with changes not considered to be caused by acute or chronic rejection Note that the Banff Diagnostic Categories form the core of the Banff Classification of Renal Allograft Pathology according the 2018 Reference Guide to the Banff Classification of Renal Allograft Pathology

CONTACTS AND LOCATIONS:
Overall Officials: Dany Anglicheau, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (1):
- Centre Hospitalier William Morey - Chalon sur Saône, Chalon-sur-Saône, Saône-et-Loire, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roufosse C, Simmonds N, Clahsen-van Groningen M, Haas M, Henriksen KJ, Horsfield C, Loupy A, Mengel M, Perkowska-Ptasinska A, Rabant M, Racusen LC, Solez K, Becker JU. A 2018 Reference Guide to the Banff Classification of Renal Allograft Pathology. Transplantation. 2018 Nov;102(11):1795-1814. doi: 10.1097/TP.0000000000002366. PMID 30028786
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Anglicheau D, Tinel C, Canaud G, Loupy A, Zuber J, Delville M, Rabate C, Scemla A, Snanoudj R, Sberro-Soussan R, Mamzer-Bruneel MF, Bererhi L, Martinez F, Timsit MO, Rabant M, Correas JM, Bienaime F, Duong JP, Helenon O, Prie D, Mejean A, Legendre C. [Renal transplantation: Procedure and early follow-up]. Nephrol Ther. 2019 Nov;15(6):469-484. doi: 10.1016/j.nephro.2019.09.001. Epub 2019 Oct 19. French. PMID 31640943
- [Background] Hermsen M, de Bel T, den Boer M, Steenbergen EJ, Kers J, Florquin S, Roelofs JJTH, Stegall MD, Alexander MP, Smith BH, Smeets B, Hilbrands LB, van der Laak JAWM. Deep Learning-Based Histopathologic Assessment of Kidney Tissue. J Am Soc Nephrol. 2019 Oct;30(10):1968-1979. doi: 10.1681/ASN.2019020144. Epub 2019 Sep 5. PMID 31488607
- [Background] Marechal E, Jaugey A, Tarris G, Paindavoine M, Seibel J, Martin L, Funes de la Vega M, Crepin T, Ducloux D, Zanetta G, Felix S, Bonnot PH, Bardet F, Cormier L, Rebibou JM, Legendre M. Automatic Evaluation of Histological Prognostic Factors Using Two Consecutive Convolutional Neural Networks on Kidney Samples. Clin J Am Soc Nephrol. 2022 Feb;17(2):260-270. doi: 10.2215/CJN.07830621. Epub 2021 Dec 3. PMID 34862241
- [Background] Jain M, Robinson BD, Salamoon B, Thouvenin O, Boccara C, Mukherjee S. Rapid evaluation of fresh ex vivo kidney tissue with full-field optical coherence tomography. J Pathol Inform. 2015 Sep 28;6:53. doi: 10.4103/2153-3539.166014. eCollection 2015. PMID 26605118